CLINICAL TRIAL: NCT03685786
Title: The Study of Autologous T Cells Expressing CD19 Chimeric Antigen Receptors Treatment of Minimal Residual Disease(MRD) of B Cell Malignancies and Then Autologous Hematopoietic Stem Cell Transplantation(Auto-HSCT)
Brief Title: CART19 Cells Treatment of MRD of B Cell Malignancies and Then Auto-HSCT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Weihong Chen06062018
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Leukemia, Lymphocytic, Acute, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell

STUDY DESIGN:
Intervention Model Description: Phase 1 Clinical Study of CD19-directed Chimeric Antigen Receptor-modified T Cells (CART19) treatment for the Patients with Minimal Residual Disease (MRD) of B Cell Malignancies and then Autologous Hematopoietic Stem Cell Transplantation(Auto-HSCT).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: CART19 cell and auto-HSCT (Experimental): CART19 cells transduced with a lentiviral vector to express anti-CD19 scFv TCRz:41BB administered by IV infusion. Auto-HSCT will be made about 6 mouths after CART19 cell is infused back to the patient.
  Interventions: Biological: CART19 cell and auto-HSCT

INTERVENTIONS:
Biological: CART19 cell and auto-HSCT — Phase 1 Clinical Study of CD19-directed Chimeric Antigen Receptor-modified T (CART19) Cells treatment for Adult Patient with Minimal Residual Disease(MRD) of B Cell Malignancies and then Autologous Hematopoietic Stem Cell Transplantation(Auto-HSCT). Subjects will receive 0.5-4 x 10^8 transduced CAR T cells as a split dose over three days as follows:Day 0, 10% fraction: 0.5-4x10^7 CART19 cells, Day 1, 30% fraction: 1.5x10^7-1.2x10^8 CART19 cells, Day 2, 60% fraction: 3x10^7-2.4x10^8 CART19 cells. Auto-HSCT will be made about 6 mouths after CART19 cell is infused back to the patient.

SUMMARY:
The clinical study of CART19 Cells treatment for MRD of B Cell Malignancies and then auto-HSCT

DETAILED DESCRIPTION:
The clinical study of the chimeric antigen receptor T cells (CART Cells) treatment for minimal residual disease(MRD) of B Cell Malignancies and then autologous hematopoietic stem cell transplantation(auto-HSCT).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CD19+, B cell Acute Lymphocytic Leukemia(B-ALL), B cell Chronic Lymphocytic Leukemia(B-CLL), B cell Lymphoma，who have 0.01%≤MRD<10% during upfront treatment 2. Patients must be within 12 months of initial B-ALL, B-CLL, B cell Lymphoma diagnosis 3. Patients must have a measurable or evaluable disease at the time of enrollment, which may include any evidence of disease including minimal residual disease detected by flow cytometry, cytogenetics, or polymerase chain reaction (PCR) analysis 4. Age 14 years to 75 years 5. Adequate organ function defined as:

1. AST and ALT ≤ 3 times upper limit of normal range for age,
2. Serum creatinine ≤ 1.6 mg/dl,
3. Direct bilirubin ≤2.0 mg/dl,
4. Adequate pulmonary function defined as ≤ grade 2 dyspnea and ≤ grade 2 hypoxia,
5. Cardiac Left Ventricle Ejection Fraction (LVEF) ≥ 40% confirmed by ECHO/MUGA. 6. Patients with CNS disease will be eligible if CNS disease is responsive to therapy 7. Expression of CD19 on leukemic blasts demonstrated by flow cytometry or immunohistochemistry of bone marrow or peripheral blood 8. Adequate performance status defined as ECOG Performance Status 0 or 1 9. Provides written informed consent 10. Subjects of reproductive potential must agree to use acceptable birth control methods, as described in protocol

Exclusion Criteria:

1. Active, uncontrolled infection
2. Active hepatitis B or hepatitis C
3. HIV Infection
4. Class III/IV cardiovascular disability according to the New York Heart Association Classification
5. Subjects with clinically apparent arrhythmia or arrhythmias who are not stable on medical management within two weeks of enrollment
6. Pregnant or nursing (lactating) women Patients with a known history or prior diagnosis of optic neuritis or other
7. immunologic or inflammatory disease affecting the central nervous system, and unrelated to leukemia or previous leukemia treatment.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-06-02 (Estimated); Study Completion 2021-09-02 (Estimated)

PRIMARY OUTCOMES:
CART19 Cells Treatment of MRD of B Cell Malignancies and Then Auto-HSCT | day 28
  The incidence of conversion of minimal residual disease (MRD) to <0.01% after CART19 therapy in patients with MRD of B Cell Malignancies during upfront treatment

CONTACTS AND LOCATIONS:
Overall Officials: Weihong Chen, M.D., Ph.D., Principal Investigator — The second people's hospital of Shenzhen, The first affiliated hospital of Shenzhen University; Xin Du, M.D., Ph.D., Principal Investigator — The second people's hospital of Shenzhen, The first affiliated hospital of Shenzhen University; Xiaochun Wan, Ph.D., Principal Investigator — Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Locations (1):
- Weihong Chen, Shenzhen, Guangdong, China

REFERENCES:
- [Derived] Zhou W, Chen W, Wan X, Luo C, Du X, Li X, Chen Q, Gao R, Zhang X, Xie M, Wang M. Benefits of Chimeric Antigen Receptor T-Cell Therapy for B-Cell Lymphoma. Front Genet. 2022 Jan 20;12:815679. doi: 10.3389/fgene.2021.815679. eCollection 2021. PMID 35126471